CLINICAL TRIAL: NCT06283550
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Evaluate the Efficacy, Safety, and Tolerability of Abrocitinib in Subjects With Moderate to Severe Chronic Hand Eczema Refractory to Corticosteroid Therapy
Brief Title: Efficacy, Safety, and Tolerability of Abrocitinib in Subjects With Moderate to Severe Chronic Hand Eczema Refractory to Corticosteroid Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INNO-6052
Record Dates: First submitted 2024-02-16; First posted 2024-02-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Chronic Hand Eczema
Keywords: abrocitinib; corticosteroid therapy; eczema; atopic dermatitis
MeSH Terms: conditions — Eczema; Dermatitis, Atopic | interventions — abrocitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Abrocitinib 200 mg (Experimental): Abrocitinib at dose 200 mg will be orally administered once daily for 32 weeks.
  Interventions: Drug: Abrocitinib 200 mg
- Abrocitinib 100 mg (Experimental): Abrocitinib at dose 100 mg will be orally administered once daily for 32 weeks.
  Interventions: Drug: Abrocitinib 100 mg
- Placebo then abrocitinib (Placebo Comparator): Placebo will be orally administered once daily for 16 weeks (Part A) then abrocitinib 200 mg will be orally administered once daily for 16 weeks (Part B).
  Interventions: Drug: Abrocitinib 200 mg; Drug: Placebo

INTERVENTIONS:
Drug: Abrocitinib 200 mg — Abrocitinib will be available in 100 mg strength tablet
  Other Names: CIBINQO
  Arms: Abrocitinib 200 mg; Placebo then abrocitinib
Drug: Abrocitinib 100 mg — Abrocitinib will be available in 100 mg strength tablet
  Other Names: CIBINQO
  Arms: Abrocitinib 100 mg
Drug: Placebo — Placebo tablet
  Other Names: Inert tablet
  Arms: Placebo then abrocitinib

SUMMARY:
This study aims to evaluate the safety, efficacy and tolerability of abrocitinib in subjects with moderate to severe chronic hand eczema, and its effects on skin biomarkers using a noninvasive method of tape stripping.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, multicenter, phase 2 study aims to evaluate the efficacy of abrocitinib in 84 adult subjects with moderate to severe chronic hand eczema, and its effects on skin biomarkers using a noninvasive method of tape stripping.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subject, 18 years of age or older, at the time of consent.
2. Subject has a history of moderate to severe CHE for at least 6 months prior to Day 1.
3. Subject has refractory hand eczema
4. Subject has moderate to severe CHE at screening and Day 1, as defined by a hand PGA of 3 or 4.
5. Contraceptive use by women of childbearing potential or their male partners during the study and until ≥ 4 weeks after the last study product administration
6. Female subject of childbearing potential has had a negative serum pregnancy test at screening and negative urine pregnancy test on Day 1.
7. Subject is willing to participate and is capable of giving informed consent.
8. Subjects must be willing to comply with all study procedures and must be available for the duration of the study.

Exclusion Criteria:

1. Subject is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study.
2. Subject has known or suspected allergic contact dermatitis of the hands and is unable to avoid exposure to the causative allergen or subjects with suspected or expected changes in irritant or allergen exposures from screening through the end of the study.
3. Subject has active skin infections of the hands.
4. Subject has a history or has current active psoriasis.
5. Subject has a history of eczema herpeticum within 12 months prior to screening, and/or a history of 2 or more episodes of eczema herpeticum in the past.
6. Subject has a history of skin disease or presence of skin condition.
7. Subject has a history of cancer prior to Day 1.
8. Subject has any clinically significant medical condition (including psychiatric condition) or physical/laboratory/vital signs abnormality.
9. Subject has a current or past medical history of conditions associated with thrombocytopenia, coagulopathy, or platelet dysfunction.
10. Subject has a current or recent clinically significant viral, bacterial, fungal, or parasitic infection.
11. Subject has a history of clinically significant heart disease.
12. Subject is ≥ 50 years old AND has a history of heart attack, other clinically significant heart problems, stroke, or blood clots (in the opinion of the investigator).
13. Presence of laboratory abnormalities at the screening visit.
14. Subject has received any marketed or investigational biological agent within 12 weeks or 5 half lives (whichever is longer) prior to Day 1.
15. Subject has used any topical treatments that could have an impact on CHE within 2 weeks prior to Day 1, including, but not limited to, topical corticosteroids, topical retinoids, crisaborole, calcineurin inhibitors, ruxolitinib, tars, bleach, bleach baths, antimicrobials, medical devices.
16. Subject has a known hypersensitivity to abrocitinib or its excipients.
17. Subject has a known history of clinically significant drug or alcohol abuse within 6 months prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in hand modified Total Lesion Symptom Score (mTLSS) | Week 16
  The mTLSS is an assessment of the severity of each of the following: erythema, scaling, lichenification/hyperkeratosis, vesicles, oedema, fissures, and pruritus/pain. Each of these are rated using a 4-point severity scale.These ratings are then added to create a total mTLSS calculated as the sum of assigned individual scores with a maximum value of 21 (most severe disease) and a minimum of 0 (no disease).

SECONDARY OUTCOMES:
Change from baseline in hand modified Total Lesion Symptom Score (mTLSS) | Weeks 2, 4 and 12
  The mTLSS is an assessment of the severity of each of the following: erythema, scaling, lichenification/hyperkeratosis, vesicles, oedema, fissures, and pruritus/pain. Each of these are rated using a 4-point severity scale.These ratings are then added to create a total mTLSS calculated as the sum of assigned individual scores with a maximum value of 21 (most severe disease) and a minimum of 0 (no disease).
Reduction from baseline in hand Physician's Global Assessment (PGA) | Weeks 2, 4, 12 and 16
  The PGA is a global assessment of the current state of the disease and will be completed specific to the hands. It is a 5-point scale of overall disease severity by rating the particular signs and symptoms of chronic hand eczema (erythema, scaling, hyperkeratosis/lichenification, vesiculation, oedema, fissures and pruritus/pain).
Change from baseline in Hand Eczema Severity Index (HECSI) | Weeks 2, 4, 12 and 16
  The HECSI scoring system incorporates both the extent and the intensity of the disease. The total sum called the HECSI score will be calculated, varying from 0 to a maximum severity score of 360 points.
Change from baseline in Extent of Disease affected with moderate to severe chronic hand eczema (CHE) | Weeks 2, 4, 12 and 16
  The Extent of Disease will be estimated by the physician as the percentage of hand area (palmar and dorsal) affected by eczema, both hands (both surface) cumulating 100%.
Patient Global Assessment (PaGA) measurements | Weeks 2, 4, 12 and 16
  Using the PaGA chart, subjects will be asked by the investigator to grade their overall change from baseline in their CHE by selecting the description which best matches their perception of treatment effect.
Change from baseline in hand Dermatology Life Quality Index (DLQI) | Weeks 2, 4, 12 and 16
  The DLQI is a simple 10-question validated questionnaire that has been used in more than 40 different skin conditions.
Change from baseline in Quality of Life in Hand Eczema Questionnaire (QOLHEQ) | Weeks 2, 4, 12 and 16
  The QOLHEQ is a disease specific instrument, thereby only assessing impairments caused by hand eczema. The QOLHEQ total-score ranges from 0-127 points.
Change from baseline in pain Numerical Rating Scale (NRS) | Weeks 2, 4, 12 and 16
  The intensity of pain related to CHE will be recorded using a NRS. Pain intensity will be evaluated by asking subjects to assign a numerical score representing of the worst intensity over the last 24 hours of their symptoms on a scale from 0 to 10, with 0 indicating no symptoms and 10 indicating the worst imaginable symptoms.
Change from baseline in itch Numerical Rating Scale (NRS) | Weeks 2, 4, 12 and 16
  The intensity of pruritus associated with CHE will be recorded using an NRS. This will be evaluated by asking subjects to assign a numerical score between 0 and 10 corresponding to their worst itching over the past 24 hours, with 0 indicating no itch and 10 indicating worst imaginable itch.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research Inc.
Locations (12):
- Canada (3):
  - INNO-6052 Site 12, Fredericton, New Brunswick
  - INNO-6052 Site 13, Cobourg, Ontario
  - INNO-6052 Site 11, Montreal, Quebec
- Poland (9):
  - INNO-6052 Site 19, Krakow
  - INNO-6052 Site 17, Lodz
  - INNO-6052 Site 21, Lublin
  - INNO-6052 Site 23, Mikołów
  - INNO-6052 Site 18, Osielsko
  - INNO-6052 Site 15, Pomorskie
  - INNO-6052 Site 20, Szczecin
  - INNO-6052 Site 16, Warsaw
  - INNO-6052 Site 22, Wroclaw

IPD SHARING:
Plan to Share IPD: No